CLINICAL TRIAL: NCT03958487
Title: Training to Deal With Distractors and With Conflicting/Problem-solving Situations: An Executive/Monitoring Treatment Protocol on Everyday Life Activities
Brief Title: An Executive/Monitoring Treatment Protocol on Everyday Life Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: María Rodríguez Bailón (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Sponsor-Investigator, María Rodríguez Bailón, Professor, University of Malaga
Organization: University of Malaga (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnosognosiaAVD2017
Record Dates: First submitted 2019-05-10; First posted 2019-05-22 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Brain Damage; Executive Dysfunction; Anosognosia
Keywords: Activities of Daily Living; Brain Injuries/rehabilitation; Generalization (Psychology); Brain Injuries/psychology; Feedback, Psychological/physiology
MeSH Terms: conditions — Brain Injuries; Agnosia

STUDY DESIGN:
Intervention Model Description: Patients with acquired brain damage and with cognitive deficits on executive/monitoring and self awareness,previously measured through neuropsychological screening
Masking Description: Patients will not be informed about the phases of the study they are in (baseline, treatment, post-treatment, follow-up)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- executive/monitoring training (Experimental): All participants will be part of the same group and their performance after treatment will be compared to their own performance prior to treatment (baseline)
  Interventions: Behavioral: Video feedback, Feedback online

INTERVENTIONS:
Behavioral: Video feedback, Feedback online — The treatment phase have 3 timepoints, 1 the patient is asked to perform an ADL alone, 2. Video feedback is administrated. This requires the participant to watch its own videotaped performance with the therapist while the therapist encourage the participant to identify errors, areas of strength, and to suggest strategies to solve errors in future sessions. 3. feedback online will be provided by the therapist on participant performance. The therapist will wait for the patient to detect and correct their error spontaneously. If the patient does not detect it, the therapist provides unspecified/specific help. This strategy is based on previous work (Schmidt, et al 2013, Ownstorth et al. 2010). The novelty of our procedure is the inclusion of distracting and conflicting/problem solving situations to be inhibited, detected and solved. Feedback will focus on these situations. The level of monitoring requirements will be adjusted to participants performance using a changing criterion design.
  Other Names: Metacognitive Training

SUMMARY:
Empirical research shows that deficits in executive/monitoring abilities (inhibition, error detection, problem solving) following acquired brain injury produce serious impact on patient's daily life performance. The authors developed an intervention method aimed at improving "on-line" error detection and correction abilities during performance of naturalistic action. Patients will be asked to complete two significant everyday activities (e.g. making a sandwich and setting the kitchen table for four people) while increasing the level of monitoring requirements as their performance improve. Monitoring requirements increased by presenting new semantically and physically related distractors and increasing the number of conflicting/problem solving situations. The treatment involves a metacognitive contextual intervention program based on providing systematic online/offline-feedback on their own performance, with emphasis on making the patient aware of how to deal with distracting/conflicting situations that were previously failed. The authors predict that errors committed and addressed through the feedback sessions (errors, actions towards distractors, failures to detect/solve conflicting situations) will be reduced on post-intervention performance compared to baseline. The authors also expect behavioral improvements to generalize to trained tasks but adding new distractors/conflicting situations or even to untrained tasks.

DETAILED DESCRIPTION:
This protocol will be applied to several acquired brain damage patients with executive/monitoring deficits. Baseline evaluation will take take around 5 sessions, The training phase will be done on 6 sessions and post-training evaluation will be completed on around 3 sessions. Each patient will be invited to be retested 8/10 weeks after completing the training, to evaluate long term effects (secondary outcome). The final number of participants enrolled in the study will depend on availability.

The authors will use a single case A-B changing criterium design: Phase A constitutes the base line. Three ADL tasks will be performed by the participant without help, two of them will be treated on phase B and the other will not be trained. Each task will be evaluated 3/4 times to obtain a robust baseline. Apart from ADL, other executive/monitoring measures will be obtained pre and post-training through neuropsychological screening.

The level of monitoring difficulty will be increasing from one training session to the next, from level 1 (2 distractors/1 conflicting situation) to level 3 (8 distractors/4 conflicting situations). Baseline and post-training performance will be evaluated at level 3.The criterion to increase the level of monitoring requirements will be adjusted to each individual depending on his/her performance on the previous level. Therefore, only if a given participant reduces on at least 75% the amount of errors from initial evaluation on the present training session he/she will be confronted with the next level of difficulty on the next session. However, if the patient doesn't reach the criterium, the same level of monitoring will be repeated and trained on the following session.

Outcomes measures (post-training phase) will be taken after completing 6 training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a chronic DCA (more than 3 months),
* Presence of cognitive deficits relative to executive/monitoring functions and/or memory evaluated by the team of professionals
* Age ≥ 18 years

Exclusion Criteria:

* Visuoperceptual deficits
* Attentional neglect
* Severe motor or perceptual alterations that impede the realization of activities of daily life
* Alterations of verbal comprehension
* Severe memory disturbances

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Number of errors on trained ADL tasks at post-training phase compared to baseline phase. | 30-45 minutes
  Target errors will be coded based on the criteria developed by Humphreys and Forde (2002). Distractor errors will be considered whenever an action is directed to a non-target object. Finally, conflicting errors will be considered whenever a conflicting situation is not detected and/or solved correctly. The authors expect to find a significant reduction on the number of errors of every category (target errors, distractor errors and conflicting errors) committed on post-training performance of trained tasks compared to baseline measures of these tasks.
Rate of old/new errors on trained ADL tasks at post-training phase. | 30-45 minutes
  The authors will codify errors as old/new, depending on whether they were already asdressed or not during the training sessions. The authors expect a reduced rate of old compared to new ones at the post-training phase.
Number of errors (target errors, distractor errors, conflicting errors) on trained ADL tasks with novel executive/monitoring requirements | 30-45 minutes
  The authors expect to find a significant reduction on the number of errors of every type (target, distractor and conflicting errors) committed at post-training performance compared to baseline even when presenting new distractors and conflicting situations that were never encountered during the training sessions. This outcome will constitute a test of near transfer.
Number of errors (target errors, distractor errors, conflicting errors) on the untrained ADL task at post-training phase compared to baseline phase | 20 minutes
  The authors expect to find a significant reduction on the number of errors o every type committed at post-training performance compared to performance at baseline, even in a task that was not trained. This outcome will constitute a test of far transfer
INECO Frontal Screening | 6-10 minutes
  Executive functions. This screening test was designed to provide health professionals with a sensitive and specific executive screening test to determine frontal dysfunction. The authors expect to find a better performance in this test at the post-training phase compared to the baseline phase. This outcome will constitute a test of far transfer.
WCPA The Weekly Calendar Planning Activity | 15-20 minutes
  This test includes the scheduling of meetings as part of a weekly planning, in total there are 10 appointments. The test provides a total error score and the ability to use problem-solving strategies.The authors expect to find a better performance in this test at the post-training phase compared to the baseline phase. This outcome will constitute a test of far transfer.
WCST Wisconsin Card Sorting Test | 10-15 min
  Evaluates the capacity of abstraction, formation of concepts and the change of cognitive strategies in response to changes that occur in environmental contingencies.The authors expect to find a better performance in this test at the post-training phase compared to the baseline phase. This outcome will constitute a test of far transfer.

SECONDARY OUTCOMES:
Measure of anticipatory awareness about own ADL performance | 3 minutes.
  Before performing every ADL task , the researcher will ask participants to evaluate how well they think they will perform (i.e. to predict the number of errors). This estimation will be compared with actual performance (number of errors committed). The difference between these two measures will constitute a measure of anticipatory awareness discrepancy, that could be positive (overestimation) or negative (underestimation). The authors expect that discrepancy in anticipatory awareness will be reduced after training compared to measures at baseline.
Measure of self awareness about own ADL performance | 3 minutes.
  After completing every ADL patients will be asked which errors they think they have committed. This estimation will be compared with actual performance (actual number of errors committed). The difference between these two measures will constitute a measure of self awareness discrepancy on their ADL performance. The Authors expect that discrepancies between patients evaluations and their actual performance will be reduced after training.
Measure of general metacognitive knowledge measured with the "Patient Competency Rating Scale" (PCRS, Prigatano, 1980). | 15 minutes.
  The PCRS is a 30-item self-report instrument which asks the subject to use a 5-point Likert scale to rate his or her degree of difficulty in a variety of tasks and functions. The subject's responses are compared to those of a significant other (a relative or therapist) who rates the subject on the identical items. Impaired self-awareness is inferred from discrepancies between the two ratings, such that the subject overestimates/underestimates his/ her abilities compared to the other informant. It includes items about competency in activities of daily living, behavioral and emotional function, cognitive abilities, and physical function.functional and cognitive competency. The authors expect that discrepancies between the patient and the caregiver will be reduced after training compared to these measures at baseline.
Follow-up of the same measures described above, taken 8/10 weeks after the end of the treatment. | 100 minutes
  The authors are interested at measuring potential long-term benefits of our intervention. To do so the authors will invite participants to be re-evaluated with most of the tests described above used at the immediate post-training phase. The authors expect to find that most improvements already present at the immediate post-training phase are still present at this follow-up time point.
Caregiver daily registration of instrumental ADL performed by the patient during the Follow-up period (during the 8/10 weeks after the end of the treatment). | 150 minutes
  The authors will include a short questionnaire for direct caregivers where they will provide information about the number of ADL performed by the patient everyday. during this time period. This information will be analyzed as a potential mediator of follow-up outcomes.

OTHER OUTCOMES:
Measures of emotional distress at post-training compared to these measures at baseline with the The Depression Anxiety Stress Scale (DASS-21, Lovibond & Lovibond, 1995) | 20 minutes
  The DASS-21, is a well-established instrument to measure symptoms of depression, anxiety and stress in both clinical and non-clinical samples of adults. It includes a total of 21 items, 7 items per subscale: depression, anxiety and stress. Patients are asked to score every item on a scale from 0 (did not apply to me at all) to 3 (applied to me very much). Sum scores are computed by adding up the scores on the items per (sub)scale and multiplying them by a factor 2. Sum scores for the total DASS-total scale thus range between 0 and 120, and those for each of the subscales may range between 0 and 42. Cut-off scores of 60 and 21 are used for the total DASS score and for the depression subscale respectively. The scale will be administrated to patients pre and post intervention in order to asses changes in emotional distress due to training. Based on previous research using similar feedback training methodology with ADL no changes are expected.

CONTACTS AND LOCATIONS:
Overall Officials: María Jesús Funes- Molina, Professor, Principal Investigator — University of Granada. Departamento de Psicología Experimental)
Locations (3):
- Spain (3):
  - Hospital Universitario Marítimo Virgen de la Victoria (Torremolinos), Málaga, España
  - Centro de Investigación Mente, Cerebro y Comportamiento (CIMCYC), Granada
  - Hospital Universitario Virgen de las Nieves. Departamento de Medicina Física y Rehabilitación., Granada

REFERENCES:
- [Derived] Salazar-Frias D, Rodriguez-Bailon M, Ricchetti G, Navarro-Egido A, de Los Santos M, Funes MJ. Training to deal with distractions and conflicting situations in activities of daily living after traumatic brain injury (TBI): Preliminary evidence from a single-case experimental design study. Neuropsychol Rehabil. 2025 May;35(4):774-809. doi: 10.1080/09602011.2024.2375495. Epub 2024 Jul 15. PMID 39010748